CLINICAL TRIAL: NCT06784284
Title: Development of a Rule for Predicting the Risk of Intracranial Hemorrhagic Injury in Elderly Patients Contacting SAMU Centre-15 for Head Trauma Following a Fall from Their Height
Brief Title: PREhospital Prediction of the Risk of Intracranial Hemorrhagic Injury in the Elderly Patient with a Fall
Acronym: PRELHIC
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: RC31/24/0518; ID RCB (Other: 2024-A02601-46)
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Intracranial Hemorrhages; Head Trauma
MeSH Terms: conditions — Intracranial Hemorrhages; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- head trauma: patient ≥ 65 years of age, calling to SAMU/centre 15 following a fall from a height (bed, chair, standing)
  Interventions: Other: Glasgow Outcome Scale -Extended (GOSE)

INTERVENTIONS:
Other: Glasgow Outcome Scale -Extended (GOSE) — Questionnaire to cotate the neurological deterioration following mild head trauma. Score from 1 to 8, the higher the number the better the outcome

SUMMARY:
Monocentric study at Toulouse University Hospital. A questionnaire collecting the elements of the study is made available to regulating physicians. The regulating doctor will take charge of the call according to the service's protocol, filling in the regulation form on the Appli-SAMU software.

A callback at D7 for patients not transferred and/or not scanned will be carried out by a clinical research associate to gather information on the neurological evolution. If, during this telephone interview, the neurological evolution is not good (GOS-E score < 7), an investigating physician will call back the patient or his trusted person/family/legal representative in order to carry out a medical assessment and propose appropriate management if necessary.

Patients who have undergone brain imaging will not be recontacted, as it has now been established that normal brain imaging performed on an emergency basis eliminates the risk of delayed cerebral hemorrhagic lesions, even in patients on anticoagulants.

DETAILED DESCRIPTION:
Monocentric study at Toulouse University Hospital. A questionnaire collecting the elements of the study is made available to regulating physicians. All callers (≥ 65 years of age) contacting center 15 for head trauma following a fall from a height are eligible. The regulating doctor will take charge of the call according to the service's protocol, filling in the regulation form on the Appli-SAMU software. He will complete the questionnaire at a later stage, once the patient has been taken into care.

A callback at D7 for patients not transferred and/or not scanned will be carried out by a clinical research associate to gather information on the neurological evolution. If, during this telephone interview, the neurological evolution is not good (GOS-E score < 7), an investigating physician will call back the patient or his trusted person/family/legal representative in order to carry out a medical assessment and propose appropriate management if necessary.

Patients who have undergone brain imaging will not be recontacted, as it has now been established that normal brain imaging performed on an emergency basis eliminates the risk of delayed cerebral hemorrhagic lesions, even in patients on anticoagulants. The medical records of these patients will be consulted by the clinical research team to collect the information required for the study.

ELIGIBILITY:
Inclusion Criteria:

* patient ≥ 65 years old
* call to the SAMU/centre 15 following a fall from a height (bed, chair, standing)
* proven or suspected head trauma

Exclusion Criteria:

* high fall kinetics (greater than 1 m or 5 steps, pedestrian knocked down)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All callers (≥ 65 years old) contacting the centre 15 for head trauma following a fall from a height
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
prediction of the risk of intracerebral haemorrhagic injury | day 7
  identify a risk of intracerebral haemorrhage with a composite criterium : identification of a traumatic haemorrhagic lesion on brain imaging performed in the emergency department or a GOS-E score (Extended Glasgow Score) of 1 to 6 at the time of the call at D7 in patients who were not transferred to an emergency department or who had not had a brain scan